CLINICAL TRIAL: NCT05773872
Title: Evaluation of Social Cognition in Patient With Type 1 or Type 2 Narcolepsy Versus Patients With Idiopathic Hypersomnia
Acronym: COGNAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: PI2022_843_0022
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Narcolepsy; Social Cognition
Keywords: Narcolepsy; social cognition
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NT1 (Experimental): type 1 narcolepsy
  Interventions: Other: Questionary
- NT2 (Experimental): type 2 narcolepsy
  Interventions: Other: Questionary
- HSI (Active Comparator): idiopathic hypersomnia
  Interventions: Other: Questionary

INTERVENTIONS:
Other: Questionary — In addition to the usual care, the patient will complete the following validated questionnaires :
  SART (Sustained Attention to Response Task), IGT (Iowa Gambling Task), UPPS (Impulsive Behaviour Scale), TAS (Toronto Alexithymia Scale), BES (Basic Empathy Scale), FRET (Facial Emotions Recognition Task), ERF-CS, MASC (Movie for the Assessment of Social Cognition)

SUMMARY:
Narcolepsy is a chronic disabling neurologic disorder mainly characterised by excessive daytime sleepiness. Type 1 narcolepsy is associated with a deficit of hypocretin in the cerebrospinal fluid responsible for the cataplexy symptom while type 2 shows a normal hypocretin level and no cataplexy. While the development of narcolepsy is independent of parental social level, narcolepsy has a significant influence on educational level, grading, social outcome, and welfare consequences. Several studies assessed global cognition efficiency, mood, and attention in narcoleptic patients but only a few specifically measured social cognition and mostly without a control group.

In a population of narcoleptics children, a severe impairment in social cognition is described for 20% of the group, contrary to 2 % for the control group. The literature also depicts some impairments in decision making, somatic and cognitive emotions responses but the emotion recognition seems to be preserved.

A better understanding of the social and cognitive aspects of narcolepsy could lead to a better treatment of the disease in its entirety, including if relevant specific cognitive behavioural therapy.

The protocol consists in a psychometric evaluation including several questionnaires in order to assess social cognition. It will be proposed to patients with type 1 or type 2 narcolepsy and patients with idiopathic hypersomnia.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (>/= 18years old)
* diagnosis of type 1 or type 2 narcolepsy or idiopathic hypersomnia
* non opposition

Exclusion Criteria:

* comorbid psychiatric or neurologic disease
* patient under 18 years old
* patient under guardianship, curators or deprived of liberty, refusal of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Mean SART score in the three groups | 2 years
  SART is Sustained Attention to Response Task. The Sustained Attention to Response Task (SART) is a computer-based go/no-go task that requires participants to withhold behavioral response to a single, infrequent target (often the digit 3) presented amongst a background of frequent non-targets (0-2, 4-9). There is evidence supporting the role of the SART as a measure of working memory, sustained attention, and impulse/inhibitory control.
Mean IGT score in the three groups | 2 years
  The Iowa gambling task (IGT) is a psychological task thought to simulate real-life decision making. Participants are presented with four virtual decks of cards on a computer screen. They are told that each deck holds cards that will either reward or penalize them, using game money. The goal of the game is to win as much money as possible. Net scores are calculated as follow: [advantageous decks (C + D) minus disadvantageous decks (A + B)] for five blocks of 20 selections.
Mean UPPS score in the three groups | 2 years
  UPPS (Impulsive Behaviour Scale). The Impulsive behavior scale (S-UPPS-P) is an instrument composed of 20 items rated on a four-point Likert scale (23): (1) disagree strongly, (2) disagree some, (3) agree some, and (4) agree strongly. Scores are presented for each of five subscales, plus a total impulsivity score. In addition to the raw scores, in order to put each subscale into the same metric, the mean is calculated for the items on each subscale, from 1 to 4, where 1 indicates that the respondent did not indorse impulsive answers, and 4 indicating a high level of self-reported impulsivity.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No